CLINICAL TRIAL: NCT00501644
Title: A Phase II Study of Chemoimmunotherapy for Patients With Potentially Platinum Sensitive Müllerian (Epithelial Ovarian, Peritoneal, or Fallopian Tube) Carcinomas
Brief Title: Chemoimmunotherapy Study for Patients With Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Bristol-Myers Squibb (Industry); InterMune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-231
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Müllerian Carcinomas; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Epithelial Ovarian; Peritoneal; Fallopian Tube; Chemoimmunotherapy; Platinum Sensitive Müllerian; Carboplatin; Paraplatin; GM-CSF; Sargramostim; Interferon Gamma; Quality of Life; QOL
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoimmunotherapy (Experimental): GM-CSF Starting dose of 400 mg injected under the skin once a day for 7 days prior to and following each course of chemotherapy + rIFN-g (Interferon Gamma) 0.1 mg injected under the skin for 2 days before and after chemotherapy (Day 5 and Day 7 of each 7-day GM-CSF cycle) + Paraplatin (Carboplatin) AUC of 5 by 1 hour IV infusion every 28 days
  Interventions: Drug: Carboplatin; Drug: GM-CSF (Sargramostim); Drug: Interferon Gamma

INTERVENTIONS:
Drug: Carboplatin — AUC of 5 by 1 hour IV infusion every 28 days.
  Other Names: Paraplatin
Drug: GM-CSF (Sargramostim) — Starting dose of 400 mg injected under the skin once a day for 7 days prior to and following each course of chemotherapy.
  Other Names: Sargramostim
Drug: Interferon Gamma — 0.1 mg injected under the skin for 2 days before and after chemotherapy (Day 5 and Day 7 of each 7-day GM-CSF cycle).
  Other Names: rIFN-g

SUMMARY:
Primary Objectives:

1. Determine response rate, time to progression, and toxicity of a schedule of carboplatin by IV (intravenous) infusion, GM-CSF and rIFN-g by SC (subcutaneous injection) in patients with potentially platinum-sensitive recurrent Müllerian carcinomas.
2. Determine whether this treatment schedule is associated with:

   1. increased levels of monocytes (>2-fold and absolute numbers 1000 cells/ml,) and of LN-DR+ DC (CD11c+ and CD123+ subsets)
   2. induction of priming and activation of MO/MA (monocytes/ macrophages), and maturation of DC (dendritic cells).
3. Determine the toxicity profile of consolidation treatment with IP (intraperitoneal) injections of rIFN-g added to carboplatin (IV) and GM-CSF (SC) for 4 doses/course.
4. Determine the effects of carboplatin plus GM-CSF and rIFN-g on quality of life in patients with platinum-sensitive Müllerian carcinomas.
5. To begin an exploration of cell surface proteins on purified activated peripheral blood and ascites monocyte/macrophages both before and after treatment with GM-CSFand rIFN-g.

DETAILED DESCRIPTION:
Carboplatin is a chemotherapy drug that is used for the treatment of ovarian cancer. GM-CSF is a protein that is used to increase the production of white blood cells. rIFN-g is a protein that stimulates cells of the immune system.

Participants will need to have pre-study blood work (about 4 teaspoons) as part of their evaluation for study entry. In addition, a chest x-ray and CT scan of the abdomen and pelvis will need to be done before any treatments.

Participants in this study will receive a frequently used dose of carboplatin by vein over 1 hour every 28 days. In addition, GM-CSF will be given for 7 days and rIFN-g will be given for 2 days before and after chemotherapy. Both drugs will be given as injections under the skin. They will be repeated with each chemotherapy course that participants receive.

GM-CSF and rIFN-g are being used to try to stimulate the immune system in the belief that this adds to the effectiveness of the chemotherapy on the tumor. During each course of chemotherapy treatment, blood samples will be taken in order to evaluate the blood count response to GM-CSF. Participants will need to remain in the Houston area beginning with the first injection of GM-CSF and for up to 9 days following the carboplatin infusion for the first course.

QOL forms will be completed at 5 separate time points during the first course of chemotherapy. Later courses will only have 2 time points for completion of the QOL forms. The completion of these forms will help researchers to evaluate the effects of the carboplatin and the 2 proteins on participants and their quality of life.

Participants will receive 3 courses of treatment (each course will include 1 treatment with carboplatin followed by 2 separate treatment cycles with GM-CSF and rIFN-g) and then be evaluated for tumor response. If the tumor is responding, 3 additional courses will be given. If after 6 courses of treatment, the tumor has completely responded and there is no evidence of the disease, then up to 4 additional courses can be given for completion of therapy. If the tumor is still responding after 6 courses but has not completely gone away, then additional courses can be given as long as the tumor is responding before completion therapy can be considered.

Completion therapy will include carboplatin given every 28 days by vein along with injections of GM-CSF under the skin before and after the chemotherapy. Injections of rIFN-g will be given directly into the abdomen through an abdominal catheter if possible. If this is not possible, then the rIFN-g will be given as injections under the skin. Participants may choose not to receive the rIFN-g through a catheter during the completion phase and can continue to receive it under the skin with the chemotherapy. A maximum of 4 additional courses can be given during this phase of the study.

Participants whose disease gets worse will be taken off the study. Participants who have intolerable side effect from the study drugs will also be taken off the study treatment. Participants will have follow up CT scans after every 3 courses of treatment. Following completion of all treatments, participants will need to return to M. D. Anderson every 3 months for follow-up exams. This will include a physical exam, blood work, and a CT scan.

This is an investigational study. A total of 65 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Müllerian carcinomas (primary epithelial ovarian, primary peritoneal, or fallopian tube) who have had a response to platinum-based chemotherapy and have a chemotherapy treatment-free interval of at least 6 months. These patients are designated potentially platinum-sensitive.
2. Measurable disease by radiological or clinical examination parameters.
3. No prior immunotherapy.
4. No concurrent steroids or radiation therapy.
5. Adequate hematological parameters (ANC >/= 1500 cells/UL, platelets >/= 100,000 cells/UL
6. Adequate renal function (serum creatinine </= 1.5 mg/dl)
7. Adequate hepatic function (serum bilirubin </= 1.5 mg/dl)
8. SGOT or SGPT </= 2.5 normal
9. Zubrod status </= 2
10. Signed informed consent
11. Patients with no more than 2 prior therapy regimens (1st line platinum and platinum reinduction will count as one)

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with brain metastases
3. Serum albumin <3 gm/dl
4. Weight loss >10% over 4 months
5. Radiation therapy to whole abdomen
6. History of clinical or EKG findings suggestive of active (within the last 6 months) heart disease
7. Patients with active autoimmune or inflammatory bowel disease
8. Patients with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
9. Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
10. Patients with prior hypersensitivity to platinum agents
11. Patients with history of other malignancy, with the exception of non-melanomatous skin cancer; unless in complete remission and off therapy for a minimum of 5 years.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Freedman, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Apte SM, Vadhan-Raj S, Cohen L, Bassett RL, Gordon IO, Levenback CF, Ramirez PT, Gallardo ST, Patenia RS, Garcia ME, Iyer RB, Freedman RS. Cytokines, GM-CSF and IFNgamma administered by priming and post-chemotherapy cycling in recurrent ovarian cancer patients receiving carboplatin. J Transl Med. 2006 Apr 7;4:16. doi: 10.1186/1479-5876-4-16. PMID 16603073
- [Result] Schmeler KM, Vadhan-Raj S, Ramirez PT, Apte SM, Cohen L, Bassett RL, Iyer RB, Wolf JK, Levenback CL, Gershenson DM, Freedman RS. A phase II study of GM-CSF and rIFN-gamma1b plus carboplatin for the treatment of recurrent, platinum-sensitive ovarian, fallopian tube and primary peritoneal cancer. Gynecol Oncol. 2009 May;113(2):210-5. doi: 10.1016/j.ygyno.2009.02.007. Epub 2009 Mar 4. PMID 19264351
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 01/07/03 to 07/25/07. All patients were recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Chemoimmunotherapy
Started | 59
Completed | 54
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemoimmunotherapy
Number analyzed (Participants) | 59
Age Continuous [Median (Full Range); unit: years] | 61 [35 to 79]
Sex/Gender, Customized [Number; unit: participants]
  Female | 59
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response
Description: Per World Health Organization (WHO) Tumor Response: Complete Response (CR), Partial Response (PR) or Progressive Disease (PD). CR defined as disappearance of all target lesions, PR as > = 30% decrease in sum of longest dimensions of target lesions with reference baseline sum longest dimensions and if CA 125 levels declined by >50%, provided target lesion size did not increase by >20% on imaging, and PD as >20% increase in sum of longest dimensions of target lesions taking as references smallest sum of longest dimensions recorded since treatment started, or appearance of 1 or > new lesions.
Time Frame: Follow up CT scans after every 3 courses of treatment and following completion of all treatments.
Population: Analysis per protocol. Of 59 participants enrolled, five (5) were not evaluable.
Measure: Number; unit: Participants
Arm/Group | Chemoimmunotherapy
Number analyzed (Participants) | 54
Participants
  Complete Response | 9
  Partial Response | 21
  Progressive Disease | 24

ADVERSE EVENTS:
Time Frame: Five years and three months
Arm/Group | Chemoimmunotherapy
Serious Adverse Events (participants affected / at risk) | 20/54
Other Adverse Events (participants affected / at risk) | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoimmunotherapy (N=54)
Neutrophil count decreased (Investigations) | 16 (16) — 12-Grade 3; 4-Grade 4
Platelet count decreased (Investigations) | 9 (9) — 9-Grade 3
Anemia (Blood and lymphatic system disorders) | 2 (2) — 2-Grade 3
Fatigue (General disorders) | 20 (20) — 16-Grade 3; 4-Grade 4
Infusion related reaction (General disorders) | 15 (15) — 15-Grade 3
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) — 10-Grade 3
Depression/Anxiety (Psychiatric disorders) | 8 (8) — 5-Grade 3; 3-Grade 4
Nausea (Gastrointestinal disorders) | 5 (5) — 5-Grade 3
Headache (Nervous system disorders) | 2 (2) — 2-Grade 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (3) — 3-Grade 3
Elevated Liver Enzymes (Investigations) | 2 (2) — 2-Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No